CLINICAL TRIAL: NCT06909513
Title: Effects of Travel Neck Pillow Usage on Cervical Comfort, Pain,Stiff Neck and Cervical Range of Motion After Thyroidectomy
Brief Title: Impact of Travel Neck Pillow Use on Neck Comfort and Mobility After Thyroidectomy
Acronym: TiNeCoM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ali BAŞGÜN, Ali BAŞGÜN, MSc, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/271; 2024/271 (Other: Erciyes Üniversitesi)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Total Thyroidectomy
Keywords: Cervical comfort; Postoperative neck pain; Neck stiffness; U-shaped Travel neck pillow; Cervical mobility; Nursing care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- U-shaped Travel Neck Pillow (Experimental): Participants in the intervention group will receive a U-shaped travel neck pillow immediately after surgery upon arrival to the ward. The pillow will be used only during rest (supine or semi-Fowler's position) for the first 24 hours postoperatively and removed before mobilization begins. After removal, assessments will include cervical comfort using the Visual Analog Scale (VAS), pain scores during neck movements (flexion, rotation, lateral flexion-excluding extension) via VAS, the McGill Pain Questionnaire for pain localization and severity, and cervical range of motion using a universal goniometer. This intervention aims to evaluate the pillow's effectiveness in reducing neck pain, stiffness, and discomfort, and improving mobility after thyroidectomy.
  Interventions: Device: U-shaped Travel Neck Pillow
- Routine Care (No Intervention): Participants in the control group will receive standard postoperative care following total thyroidectomy, without the use of a neck pillow. No additional non-pharmacological interventions will be provided. Pain management, mobilization, and other postoperative procedures will follow the hospital's routine clinical protocol. At 24 hours postoperatively, participants will be assessed for cervical comfort using the Visual Analog Scale (VAS), neck pain during movements (excluding extension) using VAS, pain localization and severity via the McGill Pain Questionnaire, and cervical range of motion using a universal goniometer. This group serves as a comparison to evaluate the effectiveness of the neck pillow intervention.

INTERVENTIONS:
Device: U-shaped Travel Neck Pillow — Participants in the intervention group will receive a U-shaped travel neck pillow immediately after surgery upon arrival to the ward. The pillow will be used only during rest (supine or semi-Fowler's position) for the first 24 hours postoperatively and removed before mobilization begins. After removal, assessments will include cervical comfort using the Visual Analog Scale (VAS), pain scores during neck movements (flexion, rotation, lateral flexion-excluding extension) via VAS, the McGill Pain Questionnaire for pain localization and severity, and cervical range of motion using a universal goniometer. This intervention aims to evaluate the pillow's effectiveness in reducing neck pain, stiffness, and discomfort, and improving mobility after thyroidectomy.
  Other Names: Travel Neck Pillow
  Arms: U-shaped Travel Neck Pillow

SUMMARY:
This study aims to evaluate the effectiveness of U-shaped travel neck pillow use in improving cervical comfort, reducing neck pain and stiffness, and enhancing cervical range of motion in adults undergoing total thyroidectomy surgery. It is the first randomized controlled trial in Turkey to examine the use of a travel neck pillow as a non-pharmacological intervention during the immediate postoperative period (day 0).

The study will be conducted at Erciyes University Gevher Nesibe Hospital between December 5, 2024 and June 5, 2025. Participants will be randomly assigned to either the pillow group or the control group. Those in the pillow group will use a U-shaped neck pillow for the first 24 hours after surgery while at rest.

Outcomes will be assessed using the Visual Analog Scale (VAS) for pain and comfort, the McGill Pain Questionnaire for pain localization and intensity, and goniometric measurements of cervical range of motion. Data will be collected preoperatively and at 24 hours postoperatively.

This study is expected to provide clinical evidence supporting the use of travel neck pillows to improve postoperative comfort and mobility, offering a simple and cost-effective nursing intervention for thyroidectomy recovery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective total thyroidectomy

Classified as ASA physical status I or II

Aged 18 years or older

No communication impairments

Willing to participate and provide informed consent

Exclusion Criteria:

* Patients with a previously diagnosed condition in the cervical spine region prior to surgery

Patients who have previously undergone thyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of Patient Comfort Using the Visual Analog Scale (VAS) | The scale was filled in the baseline
  The Visual Analog Scale (VAS) is used to measure patient comfort. It is a 10 cm (100 mm) long line that can be oriented either horizontally or vertically. On this scale, 0 indicates "extremely uncomfortable" and 100 indicates "completely comfortable." In this study, the 10 cm VAS will be used in a horizontal orientation.

OTHER OUTCOMES:
Assessment of Pain Using the Visual Analog Scale (VAS) | The scale was filled in the baseline
  The Visual Analog Scale (VAS) is a 10 cm line, drawn either horizontally or vertically, with one end labeled "no pain" and the other end labeled "worst imaginable pain." Participants are asked to mark the point on the line that best represents their level of pain. In this study, the horizontal format will be used, as it has been reported to be more reliable.
McGill Pain Questionnaire | The scale was filled in the baseline
  The McGill Pain Questionnaire (MPQ) was developed by Melzack and Torgerson in 1971 and validated in Turkish by Kuğuoğlu, Eti Aslan, and Olgun in 2003. It consists of four parts: (1) Participants indicate the pain location on a body diagram and specify whether the pain is deep (D), surface-level (Y), or both (D-Y). (2) They select descriptive words from 20 word groups that reflect the sensory, affective, and evaluative qualities of their pain. (3) The form includes items that evaluate the temporal characteristics of pain and factors that increase or reduce it. (4) Pain intensity is rated using five levels from mild to unbearable. Each response has a point value, and total scores range from 0 to 112. Higher scores indicate more severe pain.
Cervical Spine Range of Motion Assessment | The scale was filled in the baseline
  Cervical spine range of motion will be assessed using a universal goniometer, a simple protractor-like tool designed to measure joint angles. The evaluation will follow the Kendall-McCreary criteria, which define normal cervical motion as 45-65° for flexion, 45-50° for extension, 55° for rotation, and 40° for lateral flexion. To avoid compromising the surgical incision, extension will not be performed in this study. Measurements will focus on flexion, rotation, and lateral flexion.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes Üniversitesi, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided